CLINICAL TRIAL: NCT04816110
Title: Evaluation of Mineralized Plasmatic Matrix With and Without Collagen Membrane in Periimplant Bone Regeneration (Randomized Clinical Trial)
Brief Title: Evaluation of Mineralized Plasmatic Matrix With and Without Collagen Membrane in Peri-implant Bone Regeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Youmna Aboserie, Primary Investigator and oral surgeon, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPM & bone regeneration
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Horizontal Alveolar Bone Defect; Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — 1-methyl-1-piperidinomethane sulfonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mineralized plasmatic matrix with collagen membrane (Experimental)
  Interventions: Biological: mineralized plasmatic matrix with collagen membrane
- mineralized plasmatic matrix without collagen membrane (Active Comparator)
  Interventions: Biological: mineralized plasmatic matrix (MPM) without collagen membrane

INTERVENTIONS:
Biological: mineralized plasmatic matrix with collagen membrane — Two tubes of 9 ml of patient's venous blood were collected, the tubes were placed in the centrifuge machine at 2500 rpm for 12 minutes. The resultant product consists of the following two layers:
  * A yellow plasma liquid on the top of the tube.
  * Red blood cells at the bottom. - The yellow part was collected using a syringe and added to a cup that contains the bone grafting material (hydroxyapatite 20% + β-TCP 80%). The whole preparation was mixed for few seconds to obtain MPM.
  After implant placement, the buccal bone defect was grafted with MPM and covered by collagen membrane
  Arms: mineralized plasmatic matrix with collagen membrane
Biological: mineralized plasmatic matrix (MPM) without collagen membrane — Two tubes of 9 ml of patient's venous blood were collected, the tubes were placed in the centrifuge machine at 2500 rpm for 12 minutes. The resultant product consists of the following two layers:
  * A yellow plasma liquid on the top of the tube.
  * Red blood cells at the bottom. - The yellow part was collected using a syringe and added to a cup that contains the bone grafting material (hydroxyapatite 20% + β-TCP 80%). The whole preparation was mixed for few seconds to obtain MPM.
  After implant placement, the buccal bone defect was grafted with MPM.
  Arms: mineralized plasmatic matrix without collagen membrane

SUMMARY:
This study focuses on comparing the effect of MPM with or without collagen membrane on delayed implant placement in anterior maxillary aesthetic zone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missing anterior maxillary teeth and having deficient alveolar thickness.
* Good oral hygiene
* Alveolar ridge width less than 4 mm.

Exclusion Criteria:

* Medically compromised patients.
* Heavy smokers.
* Current chemotherapy or radiotherapy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | up to 1 week
  The visual analog scale was used to gauge the degree of post-operative pain with a scale from zero (lowest) to ten (highest)
Postoperative Edema | up to 1 week
  A visual descriptor analogue scale was utilized to indicate presence/ absence of edema and inflammation with a scale of zero (lowest) to 5 (highest)
Peri-implant Probing depth | up to 9 months
  Probing depth refers to the distance between the gingival margin and the bottom of the pocket. Mesial and distal pockets were measured as close as possible to contact points from the buccal aspect while facial and lingual pockets were measured at the midline of the implant. To prevent excessive tissue damage and over extension into the healthy tissue, the peri-implant sulcus depth was made with light force.
Implant stability | up to 3 months
  The implant stability was measured by Osstell®.The stability was evaluated on buccal, palatal, mesial and distal sides of the implant and the mean values of implant stability quotients ISQs were calculated. SQ, or Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.

CONTACTS AND LOCATIONS:
Overall Officials: Yomna M Abo Serie, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Moustafa El Dibany, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Gaafar N El Halawani, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt